CLINICAL TRIAL: NCT04229628
Title: Establishment of Hypertension and Diabetes Mellitus Community Management Center(HAD-COME) Project
Brief Title: Hypertension and Diabetes Mellitus Community Management Center(HAD-COME) Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019364H(R1)
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-12

CONDITIONS: Hypertension; Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This study will collect 10 mL whole blood samples from subjects at one or more study visits. The whole blood will be processed to plasma, serum and stored for testing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No special intervention — No special intervention

SUMMARY:
To develop and implement quality improvement programs for the treatment and management of hypertension and diabetes,and preventing and controlling hypertension and diabetes-related diseases in Chinese community. This program will use data collection, analysis, feedback, and process improvement to extend the use of evidence-based guidelines throughout the healthcare system and improve patient care of hypertension and diabetes in Chinese community.

DETAILED DESCRIPTION:
The aim of this project was to improving care for hypertension and diabetes mellitus in Chinese community. Study population including subjects who are hypertension and/or diabetes mellitus, of any race or ethnicity, any age.

ELIGIBILITY:
Inclusion Criteria:

* In accordance with the diagnosis of essential hypertension;
* In accordance with the diagnosis of type 2 diabetes mellitus.

Exclusion Criteria:

* Non-type 2 diabetes patients
* Secondary hypertension
* Non-hypertensive patients
* Type 1 diabetes or other types of diabetes

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Hypertension Diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of community hypertension patients receiving treatment as Chinese guideline recommended | at the time of enrollment
  Proportion of community hypertension patients receiving treatment as Chinese guideline recommended at the time of enrollment
Proportion of community diabetes mellitus patients receiving treatment as Chinese guideline recommended | at the time of enrollment
  Proportion of community diabetes mellitus patients receiving treatment as Chinese guideline recommended at the time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ying-qing, PhD, Study Director — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China